CLINICAL TRIAL: NCT05429034
Title: Effect of Acute Psychosocial Stress on Esophageal Sensitivity in Patients With Refractory Gastro-esophageal Reflux Disease
Brief Title: Effect of MIST on Esophageal Sensitivity in Patients With rGERD
Acronym: MIST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Prof Dr Jan Tack, PI, Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: S65302
Record Dates: First submitted 2021-10-20; First posted 2022-06-23 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Stress

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MIST-paradigm (Experimental): Patients assigned to the MIST paradigm arm are exposed to psychosocial stress.
  Interventions: Behavioral: MIST paradigm
- Sham-paradigm (Sham Comparator): Patients assigned to the sham paradigm are not exposed to psychosocial stress.
  Interventions: Behavioral: Sham paradigm

INTERVENTIONS:
Behavioral: MIST paradigm — Patients are exposed to psychosocial stress = receive mental arithmetic challenges, together with social evaluative threat components from the program and/or the investigator.
  Arms: MIST-paradigm
Behavioral: Sham paradigm — Patients are not exposed to psychosocial stress = threat components from the program and/or the investigator are absent
  Arms: Sham-paradigm

SUMMARY:
Effect of acute psychosocial stress on esophageal sensitivity in patients with refractory gastro-esophageal reflux disease and healthy volunteers.

DETAILED DESCRIPTION:
Gastro-esophageal reflux disease (GERD), defined as the presence of symptoms or lesions that can be attributed to the reflux of gastric contents into the esophagus, is an increasingly prevalent condition in Western societies. The most typical symptoms are heartburn and regurgitation, however GERD can also manifest itself through a variety of other esophageal and extra-esophageal symptoms (e.g. chronic cough).

GERD patients can be divided into different categories based on upper endoscopy and pH or impedance-pH (MII-pH) monitoring. In the absence of lesions (esophagitis) during upper endoscopy, a pH or MII-pH monitoring will be performed. A first subcategory are patients with true GERD, characterized by an abnormal acid exposure and a positive or negative symptom association. The second and third category are patients with reflux hypersensitivity (RHS) and functional heartburn (FH)characterized by normal acid exposure on the MII-pH monitoring and a positive and negative symptom reflux association, respectively.

The basis for symptom generation/perception in GERD patients is not yet completely understood, but different mechanisms have been proposed including esophageal hypersensitivity, in which psychosocial stress is considered as a potential factor. This was shown in a study where 64% of the participants with heartburn reported that psychological factors, such as life stress, aggravate their symptoms. Furthermore, Fass et al. observed that auditory stress exacerbated symptom perception during esophageal acid perfusion. Moreover, our group investigated the effect of intravenous corticotrophin releasing hormone (CRH) on esophageal in healthy volunteers and showed that CRH is able to increase esophageal sensitivity to mechanical distention. Nevertheless, these previously performed studies in patients have some limitations: no measurable increase in cortisol (hypothalamo-pituitary-adrenal (HPA)-axis was not affected in these studies) and patients with RHS and FH - in whom the effect of stress is hypothesized to be the most relevant - were not included.

To induce moderate psychologic stress in the current study, the Montreal Imaging Stress Task (MIST) will be used. During this protocol, participants receive mental arithmetic challenges, together with social evaluative threat components from the program and/or the investigator (sham condition: threat components from the program and/or the investigator are absent). This MIST protocol can be used when investigating the effects of perceiving and processing psychosocial stress in the human brain in functional imaging studies.

Therefore, the investigators want to investigate the relation between sensitivity to different stimuli (esophageal sensitivity) and psychosocial stress in healthy volunteers and patients (True GERD, RHS and FH).

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 to 65 years;
* Patients need to be classified as having gastroesophageal reflux disease and can be divided in three different groups (based on the Lyon consensus):

  * True GERD: Acid exposure time (AET) >6% off PPI or >80 reflux episodes on PPI
  * RHS: AET <4% off PPI or <40 reflux episodes on PPI and positive symptom association
  * FH: AET <4% off PPI or <40 reflux episodes on PPI and negative symptom association --> Result based on a measurement maximum 1 year ago.
* Subjects must be capable of understanding and be willing to provide signed and dated written voluntary informed consent before any protocol-specific screening procedures are performed.
* Being able to stop PPI intake for 10 - 14 days before the study visit.

Exclusion Criteria:

* Endoscopic signs of severe erosive esophagitis (grade C or D, Los Angeles classification) on endoscopy performed off PPI treatment in the 12 months prior to screening, or ≥ grade B when endoscopy is performed on PPI treatment;
* Systemic diseases, known to affect esophageal motility (i.e. systemic sclerosis);
* Surgery in the thorax or in the upper part of the abdomen (appendectomy and cholecystectomy are allowed);
* Significant neurological, respiratory, hepatic, renal, hematological, cardiovascular, metabolic or gastrointestinal cerebrovascular disease as judged by the investigator;
* Severe anxiety/depressive disorder (assessed with the GAD7, PHQ9 and PHQ15);
* Medication intake that affect sensitivity: anti-depressants (selective serotonin re-uptake inhibitors and tricyclic antidepressants; SSRIs and TCA and daily use of benzodiazepines);
* Pregnancy or breastfeeding;
* History of alcohol or drug abuse that would interfere with ability to comply with protocol requirements.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2024-06-22 (Estimated); Study Completion 2024-06-22 (Estimated)

PRIMARY OUTCOMES:
Esophageal mechanical sensitivity | Assessed during visit 1 at time point 75 minutes
  Change in balloon distension
Esophageal chemical sensitivity | Assessed during visit 1 at time point 180 minutes
  Change in time for reaching pain threshold

SECONDARY OUTCOMES:
Cortisol levels | every 15 minutes a saliva sample during 4.5 hours: at time points (in minutes) 0, 15, 30, 45, 60, 75, 90, 105, 120, 135, 150, 165, 180, 195, 210, 225, 240, 255, 27
  change in cortisol levels

CONTACTS AND LOCATIONS:
Locations (1):
- TARGID, Leuven, Vlaams-Brabant, Belgium